CLINICAL TRIAL: NCT06369584
Title: Efficiency and Safety of Prone Position During Extracorporeal Membrane Oxygenation in Pediatric Patients With Severe Acute Respiratory Distress Syndrome: A Multi-center Randomized Study
Brief Title: Prone Position During ECMO in Pediatric Patients With Severe ARDS
Acronym: PEPAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seventh Medical Center of PLA General Hospital (Other)
Collaborators: Gansu Provincial Maternal and Child Health Care Hospital (Other); Xian Children's Hospital (Other Government); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Henan Provincial People's Hospital (Other); Guangdong Provincial People's Hospital (Other); Shenzhen Bao'an Maternal and Child Health Hospital (Other); Zhengzhou Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEPAD
Record Dates: First submitted 2024-04-02; First posted 2024-04-17 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Acute Respiratory Distress Syndrome; Extracorporeal Membrane Oxygenation
Keywords: Extracorporeal Membrane oxygenation; pediatric acute respiratory distress syndrome; prone position ventilation
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prone position during ECMO in pediatric ARDS (Experimental): Procedure: Prone positioning The process of prone positioning requires 5-6 people, with one person acting as the commander responsible for directing and monitoring the implementation of prone positioning. The process of monitoring includes ECMO flow and vital signs. The second person is in charge of the patient's head, including endotracheal intubation, ventilator lines, and jugular ECMO cannula. The third person is responsible for femoral ECMO cannula and central venous line. The fourth to sixth individuals are responsible for rotating the patient's torso towards the side without an ECMO tube. Before initiating prone ventilation, pressure ulcer protection patches should be placed to protect areas under pressure. During ECMO support period, each patient needs to undergo at least four sessions of prone ventilation. Each session should last between 16 to 24 hours.
  Interventions: Procedure: prone position
- supine position during ECMO in pediatric ARDS (No Intervention): Procedure: Supine position Patients assigned to supine will remain in a semi-recumbent position.

INTERVENTIONS:
Procedure: prone position — The process of prone positioning requires 5-6 people, with one person acting as the commander responsible for directing and monitoring. The process of monitoring includes ECMO flow and the vital signs. The second person is in charge of the patient's head, including endotracheal intubation, ventilator lines, and jugular ECMO cannula. The third person is responsible for femoral ECMO cannula and central venous line. The fourth to sixth individuals are responsible for rotating the patient's torso towards the side without an ECMO tube. Before initiating prone ventilation, pressure ulcer protection patches should be placed on the patient's forehead, ears, anterior chest, and iliac crest to protect areas under pressure. During ECMO support period, each patient needs to undergo at least four sessions of prone ventilation until their condition improves enough to discontinue ECMO support. Each session should last between 16 to 24 hours.
  Arms: prone position during ECMO in pediatric ARDS

SUMMARY:
In 2023, the second Pediatric Acute Lung Injury Consensus Conference (PALICC-2) updated the diagnostic and management guidelines for Pediatric Acute Respiratory Distress Syndrome (PARDS). The guidelines do not provide sufficient evidence-based recommendations on whether prone positioning ventilation is necessary for severe PARDS patients. However, the effectiveness of Extracorporeal Membrane Oxygenation (ECMO) in treating severe PARDS has been fluctuating around 70% according to recent data from Extracorporeal Life Support Organization (ELSO).

In 2018, the Randomized Evaluation of Sedation Titration for Respiratory Failure (RESTORE) study group conducted a retrospective analysis and concluded that ECMO does not significantly improve survival rates for severe PARDS. However, this retrospective study mainly focused on data from North America, with significant variations in annual ECMO support cases among different centers, which may introduce bias. With advancements in ECMO technology and materials, ECMO has become safer and easier to operate. In recent years, pediatric ECMO support technology has rapidly grown in mainland China and is increasingly being widely used domestically to rescue more children promptly.

ECMO can also serve as a salvage measure for severely ARDS children who have failed conventional mechanical ventilation treatment. When optimizing ventilator parameters (titrating positive end expiratory pressure (PEEP) levels, neuromuscular blockers, prone positioning), strict fluid management alone cannot maintain satisfactory oxygenation (P/F<80mmHg or Oxygen Index (OI) >40 for over 4 hours or OI >20 for over 24 hours), initiating ECMO can achieve lung-protective ventilation strategies with ultra-low tidal volumes to minimize ventilator-associated lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Severe PARDS and meets the criteria for ECMO support, has received ECMO support for less than 48 hours.
* Informed consent obtained from the child's direct/legal guardian

Exclusion Criteria:

1. Age < 1 month or > 18 years old.
2. ECMO initiated for more than 48 hours.
3. Children who have undergone cardiopulmonary resuscitation (CPR) for more than 10 minutes before ECMO initiation without restoration of spontaneous circulation, or children undergoing extracorporeal cardiopulmonary resuscitation (ECPR).
4. Presence of irreversible brain injury or intracranial hypertension.
5. Children with irreversible lung disease awaiting lung transplantation.
6. Children with abdominal trauma or postoperative acute respiratory distress syndrome (ARDS).
7. Children in whom percutaneous cannulation cannot be performed due to unstable hemodynamics within the first 48 hours after ECMO support initiation.
8. Other contraindications for performing percutaneous cannulation.
9. Liver failure.
10. Burn area >20% body surface area (BSA).

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Day 7, Day 14, Day 30, Day 60, Day 90
  Survive means that the patient would survive without ECMO support and survival requires follow-up until at least 30 days after ECMO withdrawal. Whether the child requires long-term mechanical ventilation or home oxygen therapy after ECMO withdrawal will be considered.
  A protocolized management regarding weaning of ECMO will be applied to both groups in all involved centers.
  The planned analysis will model the risk of death.

SECONDARY OUTCOMES:
Failure of supine position | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
  The definition of failure of supine position: For patient ventilated with ECMO on supine position, when the fraction of oxygen of ECMO was set at 100% and fraction of ventilator oxygen was over 70%, saturation of the patient could not reach above 80%. This condition was defined as failure of supine position.
ECMO successful weaning rate | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
  ECMO successful weaning rate means the patient still survive for more than 48 hours after weaning from ECMO.
Total duration of ECMO Support | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
Number of ECMO-free days | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
  Number of ECMO-free days means the time for the patient to discharge from ECMO successful weaning.
Duration of mechanical ventilation days after ECMO successful weaning. | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
Duration of Pediatric Intensive Care Unit (PICU) stay. | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
Duration of hospitalization | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
Incidence of brain injury before discharge | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
  Brain injury was defined as any brain injury from imaging diagnosis or verified by EEG.
Number of days with organ failure | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
  Defined by Phoenix Sepsis Score. The Phoenix Sepsis Score ranged from 0-13, and the higher score indicates a worse prognosis.
Number of days alive without organ failure | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
  Defined by Phoenix Sepsis Score. The Phoenix Sepsis Score ranged from 0-13, and the higher score indicates a worse prognosis.
Number of ventilator assist pneumonia, bacteriemia, and cannula infection episodes | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
Number of days with hemodynamic support with catecholamines | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.
Number of days without hemodynamic support with catecholamines | Between inclusion visit (day 1) and day 60, Between inclusion visit and day 90.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Seventh medical center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Gansu Provincial Maternal and Child Health Care Hospital, Lanzhou, Gansu
  - The Second School of Clinical Medicine, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Bao'an Maternity & Child Health Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Henan Children's Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xi'an Children's Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No
All the data involved in the study should be applied for the investigator after publication.